CLINICAL TRIAL: NCT01353261
Title: Platelet Function Monitoring in Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TIMING
Record Dates: First submitted 2011-05-11; First posted 2011-05-13 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Platelet reactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Elective Cases: Patients with stable CAD undergoing PCI
- AMI Cases treated with clopidogrel: Patient with AMI undergoing PCI
- AMI Cases treated with prasugrel: Patients with AMI undergoing PCI

SUMMARY:
This study is being done to learn more about platelet reactivity (how well the small cells in the bloodstream work) in people who undergo Percutaneous coronary intervention (PCI) for stable and unstable (acute myocardial infarction) indications. Stable means you have not demonstrated any acute injury to your heart prior to your PCI; unstable means you have demonstrated some acute injury to your heart prior to your PCI. The investigators intend to determine if there is a change in platelet reactivity from the time of PCI to 30days post-PCI and does this change differ depending upon the conduction in which you present for PCI. This is going to be done with a variety of platelet reactivity assays.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old.
* Patient scheduled to undergo PCI for either stable CAD or AMI:
* Stable CAD defined as negative cardiac isoenzymes prior to the PCI as well as no resting ECG changes indicative of ACS.
* AMI defined as positive cardiac isoenzymes prior to the PCI and/or resting ECG changes indicative of ACS.

  3. Patients treated with a loading dose of clopidogrel at least 6 hours prior to the blood draw or on a maintenance dose of clopidogrel (of at least 75mg QD) for a minimum of 5 days.

Exclusion Criteria:

* Known allergies to aspirin, clopidogrel, or prasugrel
* Use of a glycoprotein (GP) IIb/IIIa inhibitor within 8 hours of the blood draw;
* Patient known to be pregnant or lactating;
* Patient with known history of bleeding diathesis or currently active bleeding;
* Platelet count <100,000/mm the day of the blood draw;
* Hematocrit <25% the day of the blood draw;
* On warfarin therapy at the time of the blood draw or the need for warfarin therapy in the subsequent month following the blood draw;
* Known blood transfusion within the preceding 10 days of the blood draw;
* Patient who has received NSAID (not including ASA) within preceding 24 hours of the blood draw;
* Patients presenting with cardiogenic shock;
* Any significant medical condition, which in the investigator's opinion may interfere with the patient's optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seventy five subjects (25 patients undergoing elective PCI for stable CAD and 50 patients undergoing urgent PCI for AMI(25 receiving clopidogrel and 25 receiving prasugrel - as determined by the treating physicians)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Platelet function | 30 days
  The primary endpoint will be whether the results of platelet function assays used to measure response to clopidogrel and prasugrel therapy is similar amongst patients with stable CAD and those with AMI undergoing PCI. On-treatment platelet reactivity will be measured using the VerifyNow P2Y12 assay.

SECONDARY OUTCOMES:
On-treatment platelet reactivity | 30 days
  A secondary endpoint will be to determine on-treatment platelet reactivity at the same time points using:
  * The vasodilator-stimulated phosphoprotein (VASP) phosphorylation assay; and/or
  * The Chrono-Log Lumi-Aggregometer, which measures platelet aggregation (via optical density or electrical impedance) in response to ADP stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States